CLINICAL TRIAL: NCT03099135
Title: A Prospective 3-Year Follow-up Study in Subjects Treated in a Preceding Phase 2 or 3 Study With a Regimen Containing Odalasvir and AL-335 With or Without Simeprevir for the Treatment of Hepatitis C Virus (HCV) Infection
Brief Title: A Long Term Follow-up Study in Participants Treated in a Preceding Phase 2 or 3 Study With a Regimen Containing Odalasvir and AL-335 With or Without Simeprevir for the Treatment of Hepatitis C Virus (HCV) Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment prematurely stopped based on decision to stop HPC program (not due to safety or efficacy results) + On 31 Jan 2018 decision to stop the study
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108301; 2016-002608-19 (EudraCT Number); 64294178HPC3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-03-30; First posted 2017-04-04 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Odalasvir and AL-335 With or Without Simeprevir (Other): Participants who completed the LPVPS (Phase 2 or Phase 3 study), in which they received a regimen containing Odalasvir and AL-335 With or Without Simeprevir for the treatment of HCV infection, and who agree to participate in this follow-up study will be assessed for durability of SVR, incidence of late viral relapse, presence and long term-persistence of resistance associated substitutions (RAS) and liver disease status.
  Interventions: Drug: No Treatment

INTERVENTIONS:
Drug: No Treatment — No treatment will be given tp participants during this follow-up study of previous phase II and Phase III in which they have received Odalavir and AL-335 with or without Simeprevir.

SUMMARY:
The main purpose of this study is to evaluate the durability of Sustained virologic response (SVR) in participants who achieved SVR at last post-therapy visit of parent studies (LPVPS) with NCT Numbers NCT02569710 and NCT02765490.

DETAILED DESCRIPTION:
This multicentre study will not provide any study treatment but collect follow-up data for up to 3 years to assess the long term durability of SVR achieved in one of the parent studies [phase 2 or 3 with AL-335 and Odalasvir (ODV) with or without Simeprevir (SMV]. In addition participants who failed to achieve an SVR in the parent study can be enrolled to assess the presence of resistance associated substitutions (RAS) and their persistance over time. It is expected that the vast majority of approximately 250 participants will enrolled in the study. Safety parameters and Liver disease status will be assessed in all participants over time.

ELIGIBILITY:
Inclusion Criteria:

* Participant was randomized to a regimen containing Odalasvir (ODV) with AL-335 with or without Simeprevir in a preceding Phase 2 or Phase 3 study (parent study)
* Participant received at least 1 dose of ODV with AL-335 with or without SMV in the parent study
* Participant has completed the last post-therapy follow-up visit of the parent study ( LPVPS) and has not passed the screening period of 6 + 3 months after the LPVPS
* Participant has signed an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Participant is currently enrolled or plans to enroll in another study with an investigational drug (including investigational vaccines) or an invasive investigational medical device between the LPVPS and Visit 6 of the present study (36 months (+/-) 4 weeks after the LPVPS of the parent study)
* Participant received antiviral or immunomodulating treatment, including therapeutic vaccines, for HCV infection between the LPVPS and the screening visit of the present study, or is planned to receive such treatment during the period of this follow-up study
* Participant is not able to adhere to the requirements of the follow-up study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Maintaining Sustained Virologic Response (SVR) Until the End of the Long-Term Follow-Up | Up to 3 years
  Participants maintained SVR if HCV RNA less than (<) lower limit of quantification (LLOQ) (Detected or Not Detected) per timepoint in this study.

SECONDARY OUTCOMES:
Percentage of Participants With Late Viral Relapse Among Participants who Achieved SVR at Last Post-Therapy Visit of Parent Study (LPVPS) | Up to 3 years
  Late viral relapse is defined as: participants who achieved SVR at LPVPS but have confirmed HCV RNA greater than or equal to (>=) LLOQ during follow-up in this study. SVR at LPVPS is defined as participants who achieved SVR12 in the parent study, and maintained HCV RNA<LLOQ until LPVPS.
Liver Disease Status in All Participants who Achieved or did not Achieve SVR at LPVPS | Up to 3 years
  Liver disease status will be evaluated using child pugh assessment score and laboratory tests including aspartate amino transferase to Platelet Ratio Index (APRI) and Metavir. Child Pugh score includes 5 clinical measures: 1) Encephalopathy grade, 2) Ascites, 3) Serum bilirubin, 4) Serum albumin, 5) Prothrombin time for assessing status of liver disease. Each measure is scored 1 to 3, with 3 indicating most severe derangement. The individual item scores will be summed to yield total score ranging from 5 to 15. Child-Pugh A (mild): 5-6 points, Child-Pugh B (moderate): 7-9 points, and Child-Pugh C (severe): 10-15 points.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- Canada (5):
  - LAIR Centre, Vancouver, British Columbia
  - Vancouver Prostate Centre, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - GI Research Institute (G.I.R.I.), Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
- New Zealand (2):
  - Auckland District Health Board, Auckland
  - Christchurch Clinical Studies Trust, Christchurch
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny im. dr Wl. Bieganskiego, Lodz
  - Hepid Diagnostyka I Terapia Tomasiewicz Kiciak Lekarze Spolka Partnerska, Lublin
  - ID Clinic, Mysłowice
- National University Hospital, Singapore, Singapore

REFERENCES:
- See also: A Prospective 3-Year Follow-up Study in Subjects Treated in a Preceding Phase 2 or 3 Study With a Regimen Containing Odalasvir and AL-335 With or Without Simeprevir for the Treatment of Hepatitis C Virus (HCV) Infection — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-002608-19/results